CLINICAL TRIAL: NCT00434993
Title: Prospective, Randomized, Multicenter Trial of Aerosolized Albuterol Versus Placebo in Acute Lung Injury
Brief Title: Drug Study of Albuterol to Treat Acute Lung Injury
Acronym: ALTA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped for futility by DSMB
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 474; N01HR056179 (NIH); HHSN268200536179C
Record Dates: First submitted 2007-01-29; First posted 2007-02-14 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Albuterol; Aerosolized; Critical Care; Ventilator
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Albuterol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albuterol Sulfate (Active Comparator)
  Interventions: Drug: Albuterol Sulfate; Procedure: Mini-Bronchoalveolar Lavage (BAL)
- Placebo (Placebo Comparator)
  Interventions: Procedure: Mini-Bronchoalveolar Lavage (BAL); Drug: Placebo

INTERVENTIONS:
Drug: Albuterol Sulfate — Albuterol sulfate, USP, solution for inhalation will be diluted as follows:
  * The full dose of 5.0 mg will be diluted into 2.0 ml of sterile normal saline solution.
  * The reduced dose of 2.5 mg will be diluted into 2.5 ml of sterile normal saline solution.
  A high-efficiency small volume jet nebulizer (SVN) powered at a flow of 8 liters/minute from a 50 psi wall oxygen flow meter will be used for continuous nebulization. The study drug will be given every 4 hours (plus or minus one hour) for ten days following randomization or until 24 hours after extubation, whichever occurs first.
  Other Names: 0.9% sodium chloride
  Arms: Albuterol Sulfate
Procedure: Mini-Bronchoalveolar Lavage (BAL) — The mini-BAL procedure involves blind specimen sampling from distal airspaces. Specimens are obtained with the Combicath (Plastimed) catheter. The procedure will be done on study days 0 and 3
  Other Names: Combicath
Drug: Placebo — Placebo aerosol will consist of 3.0 ml of identical appearing sterile 0.9 % sodium chloride without preservative.
  A high-efficiency small volume jet nebulizer (SVN) powered at a flow of 8 liters/minute from a 50 psi wall oxygen flow meter will be used for continuous nebulization (e.g.: throughout the inspiratory and expiratory cycle).
  The study drug will be given every 4 hours (plus or minus one hour) for ten days following randomization or until 24 hours after extubation, whichever occurs first.
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) and a lesser condition that occurs prior to ARDS, Acute Lung Injury (ALI), are medical conditions that occur when there is severe inflammation and increased fluids (edema) in both lungs, making it hard for the lungs to function properly. Patients with these conditions require treatment that includes the use of a breathing machine (ventilator). The purpose of this study is to find out whether giving albuterol (a drug commonly used in asthmatics) or not giving albuterol to patients with ALI or ARDS makes a difference in how long it takes for a patient to be able to breath without the ventilator.

DETAILED DESCRIPTION:
Aerosolized beta-2 agonist therapy is anticipated to diminish the formation of lung edema, enhance clearance of lung edema and decrease pulmonary inflammation in patients with acute lung injury. Because beta-2 agonists have been shown to reduce permeability induced lung injury, it is anticipated that the severity of lung injury will be reduced by aerosolized beta-2 agonist therapy. The therapy may work by enhancing resolution of pulmonary edema by upregulating alveolar epithelial fluid transport mechanisms that will in turn enhance the clearance of alveolar edema. A reduction in the severity of lung injury and the quantity of alveolar edema should result in earlier extubation and more ventilator free days, improved pulmonary oxygen uptake, and improved lung compliance.

Study design: phase II/III prospective, randomized double-blind, placebo controlled trial.

* In Phase II, patients will be treated with aerosolized albuterol 5.0 mg vs. normal saline (n=40-50)administered every 4 hours for 10 days following randomization or until 24 hours following extubation, whichever occurs first. The protocol stipulates that the 5.0 mg dose will be reduced to 2.5 mg if patients exceed defined heart rate limits.
* In Phase III, the 5.0 mg dose will be used unless there is evidence that this dose has an unacceptable safety profile or dose reductions for tachycardia occur in a large fraction of patients. In that case, a lower dose of 2.5 mg will be used.
* Patients will be followed for 90 days or until discharge from the hospital to home with unassisted breathing whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the following three criteria within a 24-hour period:

  1. Acute onset of PaO2/FiO2 less than or equal to 300 (adjustments made for altitude where appropriate)
  2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph
  3. Requirement for positive pressure ventilation via endotracheal tube
* No clinical evidence of left-sided cardiac failure to account for bilateral pulmonary infiltrates

Exclusion Criteria:

* Greater than 48 hours since all inclusion criteria are met
* Neuromuscular disease that impairs ability to ventilate without assistance, (e.g., cervical spinal cord injury at level C5 or higher spinal cord injury amyotrophic lateral sclerosis, Guillain-Barré syndrome or myasthenia gravis)
* Pregnant or breast-feeding
* Severe chronic respiratory disease (i.e., chronic hypercapnia [PaCO2 greater than 45 mmHg], chronic hypoxemia [PaO2 less than 55 mmHg on FiO2 = 0.21], hospitalization within the last 6 months for respiratory failure [PaCO2 greater than 50 mm Hg and/or PaO2 less than 55 mmHg on 0.21 FiO2], secondary polycythemia, severe pulmonary hypertension [mean PAP (pulmonary artery pressure) greater than 40 mmHg], or ventilator dependency)
* Burns over greater than 40% of total body surface area
* Cancer or other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Allogeneic bone marrow transplant within the 5 years prior to study entry
* Participant, surrogate, or physician is not committed to full support (Exception: a participant will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
* Severe chronic liver disease (Child-Pugh score of 11-15)
* Diffuse alveolar hemorrhage from vasculitis
* Morbid obesity (greater than 1kg/cm body weight.)
* Unwillingness or inability to utilize the ARDS network 6 ml / kg Predicted Body Weight (PBW) ventilation protocol
* Moribund participant and is not expected to survive 24 hours
* No intent to obtain central venous access for monitoring intravascular pressures
* Contraindication to aerosolized albuterol (see Appendix A.8 of the protocol for more information)
* Daily use (prior to study hospitalization) of inhaled beta agonist, corticosteroid, or oral leukotriene modifier
* Unwillingness of primary physician to discontinue inpatient beta agonist use
* Acute myocardial infarction or acute coronary syndrome within 30 days of study entry
* Severe congestive heart failure (see Appendix A5 of the protocol for more information)
* Participation in other experimental medication trial within 30 days of study entry with the exception of the ARDSNet pharmaconutrient nutrition trial (OMEGA)
* Heart rate greater than 85% of maximal predicted heart rate (MHR85) as calculated by MHR85 = 85% x (220-age)
* Currently receiving high frequency ventilation

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Matthay, MD, Principal Investigator — University of California, San Francisco; Roy Brower, MD, Study Chair — Johns Hopkins University
Locations (40):
- United States (40):
  - University of San Francisco-Fresno Medical Center, Fresno, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSF-Moffitt Hospital, San Francisco, California
  - UCSF-San Francisco General Hospital, San Francisco, California
  - Centura St. Anthony Central Hospital, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baton Rouge General Hospital-Blue Bonnet, Baton Rouge, Louisiana
  - Baton Rouge General Hospital-Midcity, Baton Rouge, Louisiana
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Medical Center of Louisiana, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Maryland Shock Trauma Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Rochester Methodist Hospital, Rochester, Minnesota
  - St. Mary's Hospital, Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Durham Regional Medical Center, Durham, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - Wesley Long Community Hospital, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
a deidentified database of the ALVEOLI study is available through BioLINCC

REFERENCES:
- [Derived] Brown SM, Wilson E, Presson AP, Zhang C, Dinglas VD, Greene T, Hopkins RO, Needham DM; with the National Institutes of Health NHLBI ARDS Network. Predictors of 6-month health utility outcomes in survivors of acute respiratory distress syndrome. Thorax. 2017 Apr;72(4):311-317. doi: 10.1136/thoraxjnl-2016-208560. Epub 2016 Jul 20. PMID 27440140
- [Derived] Ambrus DB, Benjamin EJ, Bajwa EK, Hibbert KA, Walkey AJ. Risk factors and outcomes associated with new-onset atrial fibrillation during acute respiratory distress syndrome. J Crit Care. 2015 Oct;30(5):994-7. doi: 10.1016/j.jcrc.2015.06.003. Epub 2015 Jun 16. PMID 26138630
- [Derived] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Matthay MA, Brower RG, Carson S, Douglas IS, Eisner M, Hite D, Holets S, Kallet RH, Liu KD, MacIntyre N, Moss M, Schoenfeld D, Steingrub J, Thompson BT. Randomized, placebo-controlled clinical trial of an aerosolized beta(2)-agonist for treatment of acute lung injury. Am J Respir Crit Care Med. 2011 Sep 1;184(5):561-8. doi: 10.1164/rccm.201012-2090OC. PMID 21562125
- See also: NHLBI Acute Respiratory Distress Syndrome Network Website — http://www.ardsnet.org
- Available data/document: Individual Participant Data Set: ARDSNet-ALTA — http://biolincc.nhlbi.nih.gov/studies/alta/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/alta/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/alta/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted with a combined Phase II/III design to enroll 1000 patients with a safety review performed after 100 subjects were enrolled and interim analysis looks at 250, 500, and 700 subjects. The first subject was entered in August 2007 and the last subject in July of 2008 when the study was stopped for futility at 282 enrolled.
Groups:
- Albuterol Sulfate: Aerosolized albuterol sulfate (5.0 mg dissolved in saline) every 4 hours
- Placebo: Preservative-free 0.9% sterile sodium chloride every 4 hours
Period: Overall Study
Arm/Group | Albuterol Sulfate | Placebo
Started | 152 | 130
Completed | 152 | 130
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol Sulfate | Placebo | Total
Number analyzed (Participants) | 152 | 130 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 111 | 100 | 211
  >=65 years | 39 | 27 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.4) | 50.9 (16.2) | 51.6 (16.2)
Gender [Count of Participants; unit: Participants]
  Female | 67 | 59 | 126
  Male | 85 | 71 | 156
Region of Enrollment [Number; unit: participants]
  United States | 152 | 130 | 282

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventilator Free Days (VFD)
Description: Ventilator-free days (VFDs) is defined as the number of days from randomization to Day 28 after achieving unassisted breathing for patients who maintained unassisted breathing for at least two consecutive calendar days. If a patient achieved unassisted breathing, subsequently required additional assisted breathing, and once again achieved unassisted breathing, we counted only the VFDs after beginning the final period of unassisted breathing. Patients who died before Day 28 were assigned zero VFDs.
Time Frame: Determined 28 days after a subject entered the study
Population: All the intent to treat patients were analyzed. Data was available on all subjects for the primary analysis only.
Measure: Mean (Standard Error); unit: days
Groups:
- Albuterol: Aerosolized albuterol sulfate (5.0 mg dissolved in saline) every 4 hours
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 152 | 130
days | 14.4 (0.9) | 16.6 (0.9)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; The trial had a statistical power of 90.7% to detect a 2.25-day increase in VFDs,assuming a SD of 10.5 days. A group sequential design was used; Test type: Superiority or Other; p = 0.087, ANCOVA — The p-value was not adjusted for multiple comparisons; Adjusted for baseline shock; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.7 to 0.3], Standard Error of Mean 1.3

2. Secondary Outcome: Mortality Prior to Hospital Discharge With Unassisted Breathing to Day 60
Description: Success for this efficacy variable was defined as being alive on study day 60 or having been discharged alive off mechanical ventilation from the study hospital (or subsequent hospital) to the subject's original place of residence. Those subjects alive in hospital at day 60 were considered to have survived.
Time Frame: Determined 60 days after a subject entered the study
Population: Intent to treat population.
Measure: Number; unit: percentage of participants who died
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 152 | 130
percentage of participants who died | 23.0 | 17.7
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.302, Regression, Logistic — The p-value was not adjusted for multiple comparisons; Adjusted for baseline shock; Risk Difference (RD) = 5.3, 95% CI 2-sided [-4.0 to 14.7]

3. Secondary Outcome: Mortality Prior to Hospital Discharge With Unassisted Breathing to Day 90
Description: Success for this efficacy variable was defined as being alive on study day 90 or having been discharged alive off mechanical ventilation from the study hospital (or subsequent hospital) to the subject's original place of residence. Those participants who still remained in the hospital at 90 days after randomization were considered to have survived.
Time Frame: Determined 90 days after a subject entered the study
Population: Intent to treat.
Measure: Number; unit: percentage of participants who died
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 152 | 130
percentage of participants who died | 24.3 | 18.5
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.261, Regression, Logistic — The p-value was not adjusted for multiple comparisons; Adjusted for baseline shock; Risk Difference (RD) = 5.9, 95% CI 2-sided [-3.7 to 15.4]

4. Secondary Outcome: Number of ICU-free Days at 28 Days After Randomization
Description: ICU (intensive care unit)-free days was defined as the number of days a subject was out of the ICU during study hospitalization from date of randomization up to study day 28. All incidences of ICU admission and discharge during the study hospitalization were captured. Any portion of a calendar day that a subject was in the ICU was counted as an ICU day.
Time Frame: Determined 28 days after a subject entered the study
Population: Intent to treat.
Measure: Mean (Standard Error); unit: days
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 152 | 130
days | 13.5 (0.8) | 16.2 (0.8)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.023, ANCOVA — The p-value was not adjusted for multiple comparisons; Adjusted for baseline shock; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.9 to -0.4]

5. Secondary Outcome: Number of Organ Failure-free Days at Day 28 Following Randomization
Description: Subjects were followed for development of organ failures from date of randomization to hospital discharge or study day 28, whichever was first. Organ failure was defined as present on any calendar day when the most abnormal vital signs or clinically available lab value met the definition of clinically significant organ failure according to the Brussels Organ Failure Table. Each day a patient was alive and free of a given clinically significant organ failure was scored as a failure-free day. The worst value for a calendar day was captured (lowest systolic BP, platelet count and highest creatinine and bilirubin values). Specific definitions of organ failure were: cardiovascular-systolic BP less than or equal to 90 mmHg or on a vasopressor; coagulation-platelet count less than or equal to 80 x 1000/mm3; Renal-creatinine less than or equal to 2.0 mg/dL; Hepatic-bilirubin less than or equal to 2.0 mg/dL.
Time Frame: Daily from baseline to study day 28
Population: Intent to treat.
Measure: Mean (Standard Error); unit: days
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 152 | 130
days | 14.2 (0.9) | 15.9 (1.0)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.226, ANCOVA — The p-value was not adjusted for multiple comparisons; Adjusted for baseline shock; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.3 to 0.9]

6. Secondary Outcome: Ventilator Free Days to Day 28 in the Subset of Participants With ARDS
Description: Difference in the main outcome Ventilator Free Days to study day 28 was calculated for the subset of patients with ARDS (defined as a PaO2/FiO2 ratio of less than or equal to 200). P/F ratio is an index of the effectiveness of arterial oxygenation that corresponds to the ratio of partial pressure of arterial O2 to the fraction of inspired O2. VFD to Day 28 is defined as the number of days from the end of ventilation to day 28 in patients who maintained unassisted breathing for at least two consecutive calendar days. Patients who died before day 28 were assigned a VFD count of zero. If a patient returned to assisted breathing, subsequently required assisted breathing, and once again achieved unassisted breathing, only the VFDs after beginning the final period of unassisted breathing were counted. An increase in the number of VFDs was considered a positive result.
Time Frame: Determined 28 days after a subject entered the study
Population: Patients meeting the criteria for ARDS (pre-randomization PaO2/FiO2 ratio less than or equal to 200) were selected for this subset.
Measure: Mean (Standard Error); unit: days
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 106 | 86
days | 14.5 (1.1) [14 to 22] | 16.8 (1.0) [19 to 23]
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.130, ANCOVA; Adjusted for baseline shock; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-5.3 to 0.6]

7. Secondary Outcome: Hospital Mortality to Day 60 in the Subset of Participants With ARDS
Description: Difference in the main outcome mortality to study day 60 was calculated for the subset of patients with ARDS (defined as a PaO2/FiO2 ratio of less than or equal to 200) prior to randomization. P/F ratio is an index of the effectiveness of arterial oxygenation that corresponds to the ratio of partial pressure of arterial O2 to the fraction of inspired O2.
Time Frame: Determined 60 days after a subject entered the study
Population: as for outcome 6
Measure: Number; unit: percentage of participants who died
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 106 | 86
percentage of participants who died | 24.5 | 16.3
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.176, Regression, Logistic; Adjusted for baseline shock; Risk Difference (RD) = 8.2, 95% CI 2-sided [-3.1 to 19.6]

8. Secondary Outcome: Ventilator Free Days to Day 28 in the Subset of Patients With Baseline Shock
Description: Difference in the main outcome Ventilator Free Days to study day 28 was calculated for the subset of patients who were in shock at the time of randomization. Shock was defined as mean arterial pressure<60 or the need for vasopressors (except dopamine <6 ug/kg/min).
Time Frame: Determined 28 days after a subject entered the study
Population: Patients with protocol defined shock (mean arterial pressure<60 or need for vasopressors except dopamine < 6ug/kg/min) at the time of study entry.
Measure: Mean (Standard Error); unit: days
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 68 | 55
days | 10.0 (1.3) [0 to 18] | 13.9 (1.4) [10 to 22]
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.048, ANCOVA; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-7.8 to -0.0]

9. Secondary Outcome: Hospital Mortality up to Day 60 in Subjects With Baseline Shock
Description: Difference in the main outcome hospital mortality to study day 60 was calculated for the subset of patients who were in shock at the time of randomization. Shock was defined as mean arterial pressure<60 or the need for vasopressors (except dopamine <6 ug/kg/min).
Time Frame: Determined 60 days after a subject entered the study
Population: as for outcome 8
Measure: Number; unit: percentage of participants who died
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 68 | 55
percentage of participants who died | 36.8 | 27.3
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Test type: Superiority or Other; p = 0.265, Regression, Logistic; Risk Difference (RD) = 9.5, 95% CI 2-sided [-6.9 to 25.9]

10. Secondary Outcome: Plasma Levels of IL-6 and IL-8 on Study Day 3
Description: Biologic end-points were selected that would provide mechanistic insight into how albuterol improved lung function. Concentrations of two proinflammatory cytokines, interleukin 6 and 8 (IL-6 and IL-8), were measured. Plasma was collected and cytokine levels were measured at baseline and 3 days after randomization. IL-6 and IL-8 levels were normalized using log transformation. Wilcoxon's test was used to compare mean log-transformed interleukin levels per day and a mixed-effects model was fit to compare the slopes.
Time Frame: Measured at baseline and 3 days after randomization
Population: Not all subjects had available data for secondary analyses and therefor the numbers will be less than the 152 (active) and 130 (placebo) arms.
Measure: Log Mean (Standard Deviation); unit: pg/ml
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 127 | 110
pg/ml
  IL6 | 1.9 (0.6) | 1.8 (0.7)
  IL8 | 1.7 (0.5) | 1.7 (0.5)

ADVERSE EVENTS:
Arm/Group | Albuterol Sulfate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/152 | 1/130
Other Adverse Events (participants affected / at risk) | 21/152 | 15/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol Sulfate (N=152) | Placebo (N=130)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol Sulfate (N=152) | Placebo (N=130)
Arrhythmias (clinically important) (Cardiac disorders) | 15 (29) | 8 (11)
Hypokalemia (Metabolism and nutrition disorders) | 8 (12) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No